CLINICAL TRIAL: NCT02963142
Title: A Molecular Toolkit for the Microbial Investigation of Severe Community Acquired Pneumonia (S-CAP Study)
Brief Title: A Molecular Toolkit for the Microbial Investigation of Severe Community Acquired Pneumonia
Acronym: S-CAP
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: SCAP2016
Record Dates: First submitted 2016-10-27; First posted 2016-11-15 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2018-08

CONDITIONS: Community Acquired Pneumonia; Respiration Failure; Pneumonia
Keywords: Intensive care; Extra-corporeal membrane oxygenation (ECMO); Severe Respiratory Infections; Sequencing; Metagenome; Diagnosis
MeSH Terms: conditions — Community-Acquired Pneumonia; Respiratory Insufficiency; Pneumonia; Respiratory Tract Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, bronchoalveolar lavage,nose and throat swab and oropharyngeal swabs.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- SCAP requiring ECMO: Patients diagnosed with severe respiratory failure due to community acquired pneumonia that require extra-corporeal membrane oxygenation and a routine bronchoscopy for clinical purposes.
  Molecular laboratory techniques will be applied to residual respiratory tract samples including bronchoalveolar lavage and non-directed bronchoalveolar lavage. Comparisons will be made to conventional diagnostic tests used in the diagnosis of community acquired pneumonia.
- SCAP requiring ITU support: Patients diagnosed with severe respiratory failure due to community acquired pneumonia that require intensive care support and undergo a routine bronchoscopy for clinical purposes.
  Molecular laboratory techniques will be applied to residual respiratory tract samples including bronchoalveolar lavage and non-directed bronchoalveolar lavage. Comparisons will be made to conventional diagnostic tests used in the diagnosis of community acquired pneumonia.
- Healthy controls: Healthy volunteers who undergo bronchoscopy as part of a designated research bronchoscopy list.
  Molecular laboratory techniques will be applied to bronchoalveolar lavage samples.

SUMMARY:
Severe community acquired pneumonia is common and associated with high mortality. Conventional microbiological diagnostics identify pathogens in approximately half of cases, which is inadequate for both clinical and epidemiological purposes. This study applies next-generation sequencing based metagenomic techniques to patients with extremely severe community acquired pneumonia, to investigate the microbiome of severe community acquired pneumonia and evaluate metagenomic approaches as diagnostic tools.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or over
* Admitted to a participating severe respiratory failure centre or ICU
* Admitted due to community acquired pneumonia (CAP) according to clinical and radiological criteria
* Tracheal intubation, receiving mechanical ventilation +/- ECMO
* Requires bronchoscopy as part of routine diagnostic care plan
* Bronchoscopy takes place within 72 hours of first admission to hospital

Exclusion Criteria:

* Any current or previous condition/circumstance that, in the opinion of the investigator or study nurse, may put the individual at risk if participating
* Patients receiving end of life care
* Hospitalisation within the previous 28 days (not including pre-ECMO hospitalisation for ECMO patients)
* Consent or assent not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults admitted to Extra-Corporeal Membrane Oxygenation (ECMO) and Intensive Care Units (ICU) centres in England for severe community-acquired pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Detection of pathogens by metagenomic sequencing applied to bronchoalveolar lavage samples | 28 days (From time of enrollment up until end of inclusion)
  The proportion of pathogen genome that can be detected in bronchial lavage samples detected by the proportion of the sequenced nucleic acid which is pathogen derived and the proportion of the pathogen genome which be reconstructed.

SECONDARY OUTCOMES:
Metagenomic detection of pathogen genomes compared to the results of conventional diagnostic techniques | 28 days (From time of enrollment up until end of inclusion)
  Metagenomic sequencing data obtained will be compared to results obtained from conventional diagnostic tests undertaken as part of the participant's routine clinical care. Data will be used to evaluate the ability of each technique to detect any pathogens found.
  The conventional microbiological tests that will be used for comparison include those undertaken as part of the participants routine clinical care and will include urinary antigen tests (Pneumococcal and Leigonella); blood, sputum and bronchial lavage culture including polymerase chain reaction (PCR) for Legionella spp, Mycoplasma pneumoniae and Chlamydophila pneumoniae and respiratory viral PCR multiplex assays. The results of serological tests and PCR for Influenza A &B from nose and throat swabs will also be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ajit Lalvani, MBBS,MRCP,FRCP, Study Chair — Imperial College London
Locations (1):
- Ajit Lalvani, Paddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided